CLINICAL TRIAL: NCT00476918
Title: Dosage Dependency of Intravitreal Triamcinolone Acetonide for Treatment of Diabetic Macular Edema
Brief Title: Intravitreal Triamcinolone Acetonide for Diabetic Macular Edema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 21091968; Insurance no.: 20-770-968594
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: diabetic macular edema; triamcinolone acetonide; intravitreal; steroid
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Intravitreal Injections; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Intravitreal injection (triamcinolone acetonide)

SUMMARY:
Efficacy duration of triamcinolone acetonide (steroid) for treatment of diabetic macular edema. Furthermore, dosage dependency of triamcinolone acetonide comparing a high dosage versus a low dosage.

DETAILED DESCRIPTION:
Patients with diabetic retinopathy suffer from visual acuity loss caused by diabetic macular edema. Intravitreal injected Triamcinolone Acetonide (steroid) reduces macular edema and increases visual acuity. The duration of its effect is however limited. Therefore, several injections are necessary.

In this study a dosage dependency of triamcinolone acetonide (high dosage vs low dosage) is performed. The primary outcome parameters are the number of treatments and the efficacy of each injection.

ELIGIBILITY:
Inclusion Criteria:

* diabetic macular edema and visual acuity between 20/200 and 20/40 age over 18 years

Exclusion Criteria:

* recent treatment with laser photocoagulation or intravitreal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-07; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity, no of treatments, duration of efficacy | 12 months

SECONDARY OUTCOMES:
intraocular pressure, retinal thickness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jost Jonas, PhD MD, Study Director — Dep of Ophthalmology, University of Mannheim
Locations (1):
- Dep of Ophthalmology, University of Mannheim, Mannheim, Germany